CLINICAL TRIAL: NCT04017052
Title: Application of a TBE-Vaccine in Obese Persons
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Ursula Wiedermann, Head of Institute of Specific Prophylaxis and Tropical Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TBE_obesity_1.1
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Tick Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — FSME-IMMUN vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Booster vaccination (Other): Intervention = one i. m. TBE booster vaccination (FSME-Immun) at visit 1.
  Interventions: Drug: FSME-IMMUN Vaccine

INTERVENTIONS:
Drug: FSME-IMMUN Vaccine — Booster with TBE vaccine (i.m.) FSME Immun

SUMMARY:
Obese people have an altered immune responsiveness. The present study investigates whether this influences immune responses to booster vaccinations (i. e. booster vaccination with TBE vaccine "FSME Immun") and if a modification of vaccination schedules is needed.

Obese adults (BMI >30) >18 - 60 years are compared with adults with normal weight (BMI <25) concerning TBE-NT- antibody titers, TBE- NT antibody titer course and cellular immunity. Metabolic parameters and sexual hormones will be tested and compared as well.

DETAILED DESCRIPTION:
Obese people have an altered immune responsiveness. Studies have shown that obesity has a direct effect on the immune system and leads to immunosuppression, which leads to a susceptibility to infection.We investigate whether this influences immune responses to booster vaccinations (i. e. booster vaccination with TBE vaccine "FSME Immun") and if a modification of vaccination schedules is needed.

The investigators will test and compare the humoral and cellular immune response of obese persons (BMI>30) and persons with normal weight (BMI<25) before and after a booster with FSME Immun.

The aim of the study is to clarify if a modification of vaccination schedules or a change of booster intervals is necessary for obese people. Furthermore this study will increase our understanding of the influence of obesity on different components of the immune system, as well as on the quality and quantity of the immune responses.

At Screening (visit 1) demographic parameters (age, gender, weight, BMI, waist/hip-ratio) will be recorded and metabolic parameters (Cholesterol, Triglycerides, HDL, LDL, Apolipoproteine, Lp(a), Glucose, Fructosamin, Leptin, Leptinreceptor on T- and B-cells (PCR), Insulin, high-sensitive CRP) and sex hormones (Testosterone, Estrogen, Progesteron, FSH, LH) will be tested. At visit 3 some metabolic parameters (Cholesterol, Triglycerides, HDL, Glucose, Fructosamin, Insulin und high-sensitive CRP) will be tested again. All parameters will be compared and correlated with humoral and cellular immune responses.

Immunglobulins: IgG, IgE, IgD, IgM, IgA will be tested at visit 1-4.

TBE antibody titers (NT) will be tested and titer course will be evaluated at visit 1-5.

At visit 1 und 2, isolation of PBMC (Peripheral Blood Mononuclear Cells) with Ficoll gradient will be carried out and the following tests will be performed:

1. Cytokine concentrations will be measured after re-stimulating the PBMC with TBE-Antigen. Duration of stimulaton: 48h; Detection with Luminex platform/ELISA: IL-2, IFNgamma, IL-10, TNF-alpha und IL-6
2. Flow cytometry: Characterization of different lymphocyte-subpopulations with antibody-panels (CD surface markers: CD19, CD3, IgD, IgM, IgG, IgA, CD10, CD27, CD127, CCR4, CD8, CD4, CD28, CD31, CD38, CCR7, CD45RA, CD25, CD24, CD38 und FOXP3).

Serious adverse events and adverse events will be recorded at all visits

All participants will be tested again at V5, performing TBE-Neutralisation-Test three years after the booster vaccination for analysis of longterm immunogenicity. Demographic parameters will be recorded again.

Participants who are not protected against TBE for another year, three years after the booster vaccination at V5 (NT <20), will receive a booster vaccination for free.

V1 day 0, V2 day 7+3,V3 1 month +/-7 days, V4 6 months +/-14d V5 36 months+/- 1 month V6 only if TBE NT<20

ELIGIBILITY:
main Inclusion Criteria:

* willingness to sign written informed consent form
* completed primary TBE immunization and at least 1 booster vaccination
* participants of both sexes between 18 and 60 years of age

main Exclusion Criteria:

* age < 18 and > 60 years
* BMI 25-30
* previous TBE infection
* pregnancy or breast feeding
* acute infection on day of inclusion (day 0) or at visit 5 (36 months), body temperature > 37,9°C
* concomitant medications: systemic cortison therapy, chemotherapy, immunotherapy (allergy) immunsuppressive therapy 4 weeks prior or during the study
* administration of other vaccines 4 weeks before/after day 0
* planned surgery within 2 weeks before/after TBE booster
* any contraindication to administration of FSME-Immun® vaccine according to manufacturer's instructions
* malignant diseases within 5 years prior to the study
* autoimmune diseases
* kidney insufficiency, dialysis
* drug addiction
* plasma donor
* receipt of blood transfusions or immunoglobulins within 3 months prior to study entry / within 3 months prior to visit 5
* Severe disease with hospitalization or surgery 3 months before or during the study
* participation in a clinical trial simultaneously to visit 1-4 with receipt of vaccination and/or investigational product within one month before booster

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2020-02-07 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Humoral immunity (TBE NT) | 1 month +/- 7 days after booster (v3)
  Humoral immunity tested with TBE Neutralisation test- Neutralizing antibody titer against TBE

SECONDARY OUTCOMES:
TBE-NT titer course | before booster at day 0 at all visits until 3 years after booster vaccination at V5 (36 months+/-1 month)
  TBE-NT titer course evaluation
Cellular immune response with flow cytometry | evaluated before (V1 day 0) and 1 week after booster vaccination (V2 day 7+3d)
  Cellular immune response:
  Characterisation of lymphocyte sub-population with flow cytometry: detection of CD surface markers of lymphocytes with antibody panels - CD19, CD3, IgD, IgM, IgG, IgA, CD10, CD27, CD127, CCR4, CD8, CD4, CD28, CD31, CD38, CCR7, CD45RA, CD25, CD24, CD38 und FOXP3
Measurement of Cytokines with Luminex platform/ELISA | evaluated before (V1 day 0) and 1 week after booster vaccination (V2 day 7+3d)
  Measurement of cytokines IL-2, IFNgamma, IL-10, TNF-alpha und IL-6 in supernatants of PBMC cultures re-stimulated with TBE antigen; duration of stimulation: 48h.
  Measurement with Luminex Platform/ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann-Schmidt, MD, PhD, Principal Investigator — Medical University of Vienna , ISPTM
Locations (1):
- Medical University Vienna, Institute of Specific Prophylaxis and Tropical Medicine, Vienna, Austria

REFERENCES:
- [Derived] Garner-Spitzer E, Poellabauer EM, Wagner A, Guzek A, Zwazl I, Seidl-Friedrich C, Binder CJ, Stiasny K, Kundi M, Wiedermann U. Obesity and Sex Affect the Immune Responses to Tick-Borne Encephalitis Booster Vaccination. Front Immunol. 2020 May 27;11:860. doi: 10.3389/fimmu.2020.00860. eCollection 2020. PMID 32528467